CLINICAL TRIAL: NCT02470676
Title: Cervical Pessary vs. Vaginal Progesterone in Preventing Preterm Birth Among Women Presenting With Short Cervix: An Open-label Randomized Controlled Trial
Brief Title: Cervical Pessary vs Vaginal Progesterone in Preventing Preterm Birth Among Women Presenting With Short Cervix: An Open-label Randomized Controlled Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0096-14-HYMC
Record Dates: First submitted 2015-06-04; First posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Preterm Birth; Short Cervix
MeSH Terms: conditions — Premature Birth | interventions — Pessaries; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone (Active Comparator): 200 mg daily of vaginal progesterone suppositories (Utrogestan)
  Interventions: Drug: Progesterone
- Progesterone plus Experimental device (Experimental): Experimental device + 200 mg daily progesterone vaginal suppositories (Utrogestan)
  Interventions: Device: Pessary

INTERVENTIONS:
Device: Pessary — Two optional pessary sizes with the following dimensions: 65/17/35 or 70/17/35 and 200 mg daily progesterone vaginal suppositories (Utrogestan)
  Arms: Progesterone plus Experimental device
Drug: Progesterone — 200 mg daily of vaginal progesterone suppositories (Utrogestan)
  Arms: Progesterone

SUMMARY:
The purpose of this randomized control trial is to determine whether cervical pessary plus vaginal progesterone is superior to vaginal progesterone alone in decreasing preterm delivery rate, and improving perinatal outcome, among women presenting with an asymptomatic mid-pregnancy short cervix, in singleton and twin gestations.

All women with singleton or twin pregnancies undergoing routine ultrasonography up to 24 completed weeks of gestation (for examination of fetal anatomy and growth) and diagnosed with cervical length of ≤25 mm in singleton, or ≤38 mm in twins, will be invited to participate in the clinical trial.

Women who meet eligible criteria will be invited to participate in the clinical trial.

Women will be randomly assigned into one of the following groups: group A (vaginal progesterone) or group B (vaginal progesterone + pessary).

Follow-up visits for ultrasound assessment of fetal growth and cervical length will be carried out every two weeks until 37 weeks of gestation.

DETAILED DESCRIPTION:
Preterm birth represents a major challenge to obstetricians as well as healthcare policy makers. It is a leading cause of perinatal morbidity and mortality among singleton and multiple pregnancies. In the USA, the frequency of of preterm births (<37 completed weeks of gestation) is 10-13% in singleton pregnancies, and 57% in twins and these rate have not substantially changed in the last decade.

A short cervix (<25 mm) measured by vaginal ultrasonography during mid pregnancy (18-24 weeks of gestation) is a powerful predictor of spontaneous preterm birth (PTB). The relative risk for PTB increases as the cervical length decreases.

The two most studied treatment options in cases of short cervix at mid pregnancy are vaginal progesterone preparations, and cervical cerclage. Vaginal progesterone, given either as 90 mg gel or 200 mg suppository, was repeatedly shown to significantly reduce PTB rates and perinatal morbidity and mortality in women found to have a short cervix (20 mm or less) at 24 weeks gestation.

Progesterone were proven ineffective for the prevention of preterm birth in cases of multiple gestations, present preterm labor, or preterm premature rupture of membranes.

Cerclage may be considered an alternative for vaginal progesterone only in women with history of PTB that are found to have a short cervix in the present pregnancy (cervical length <25 mm before 24 weeks of gestation). According to a recently published indirect meta-analysis, vaginal progesterone and cerclage are equally efficacious in the prevention of PTB in women with a singleton gestation, mid trimester sonographic short cervix, and a history of previous preterm birth.

Unfortunately, vaginal progesterone and cervical cerclage were not proven effective for the prevention of PTB in twin gestations. Moreover, cervical cerclage in this context may even lead to worse outcome compared to conservative treatment. Additionally, in contrast to singleton pregnancies, neither vaginal progesterone nor injections of 17alpha-hydroxyl-progesterone caproate prevented neonatal morbidity or preterm birth in multiple pregnancies. One meta-analysis suggested that vaginal progesterone for mid trimester short cervix in twin gestation may improve neonatal outcome without prolonging the pregnancy.

Cervical Pessary is a renovated method, currently being studied for its clinical advantages over the existing available treatments in the context of midtrimester asymptomatic short cervix in singleton and twin gestation.

The largest multicenter randomized controlled trial (RCT) on pessary use in selected women screened by Trans Vaginal Sonography (TVS) excluded women who had one of the following: a known major fetal anomaly, painful regular uterine contractions, active vaginal bleeding, ruptured membrane, placenta previa, or a history of cone biopsy or cervical cerclage in situ. The conclusion of this study was that in women with a short cervical length (>25mm) between 18-22 weeks, the use of cervical pessary significantly prolonged pregnancy and reduced the rate of poor neonatal outcome compared with control, untreated patients. A second, and smaller, RCT failed to corroborate the findings previously described. In this study, the mean gestational age at delivery was 38.1 weeks in the pessary group compared to 37.8 weeks in the expectant management group, with no significant differences in the rates of delivery before 28, 34 or 37 weeks of gestation.

Currently, no published RCT compared the efficacy of the cervical pessary with that of cerclage or progestogens for short cervix in singletons or twins. A retrospective comparison between the methods has shown no significant differences in the rates of perinatal loss, neonatal morbidity or PTB for singleton pregnancies (apart from higher rate of PTB at <34 weeks' gestation in the vaginal progesterone vs the pessary group).

In 2003, the first case control study in twin pregnancies and cervical pessary was conducted. Twenty-three women with short cervical length (<25 mm) prior to 24 weeks of gestation were treated with pessary and matched with 23 controls. The mean gestational age at delivery was 35+6 weeks in the pessary group and 33+2 weeks in the control group (p value=0.02).

A large RCT published in 2013 included 403 women with twin pregnancies who were randomized to either prophylactic pessary or expectant management. Women with all cervical length were included. The authors concluded that prophylactic use of pessary in unselected twin pregnancies did not prolong pregnancy or reduce poor perinatal outcome. However, in a sub group analysis of women with a cervical length less than 38 mm (<25th percentile), a significantly lower incidence of poor neonatal outcomes, delivery before 32 weeks, and neonatal mortality was found in the pessary group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed to be pregnant at up to 24+0 weeks of gestation, with a cervical length measurement of ≤25 mm with a singleton pregnancy, or ≤38 mm in twins pregnancy.
* Does not meet with maternal/fetal/membrane/placental factors detailed in the exclusion criteria.
* Willingness to comply with the protocol for the duration of the study.
* Have signed an informed consent.

Exclusion Criteria:

* Fetal factors: major fetal abnormalities, death of one or both of the fetuses, twins- twin-to-twin transfusion syndrome, and severe growth retardation.
* Maternal factors: prophylactic cervical cerclage in situ, painful regular uterine contractions, active labor, active vaginal bleeding, maternal age under 18, uterine abnormalities (i.e. two cervices), and severe uterine prolapse.
* Membranes and placental factors: placenta previa, ruptured membranes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
preterm birth before 34 weeks of gestation rate in singleton pregnancies | up to 20 weeks from recruitment
preterm birth before 32 weeks of gestation rate in twin pregnancies | up to 20 weeks from recruitment

SECONDARY OUTCOMES:
Other preterm birth age before 34, 28 weeks in twin pregnancies | up to 20 weeks from recruitment
Neonatal/perinatal complications rate | up to 20 weeks from recruitment
  Respiratory Distress Syndrome (RDS), necrotizing enterocolitis, intraventricular hemorrhage, proven neonatal sepsis, retinopathy of prematurity, bronchopulmonary dysplasia, periventricular leukomalacia, fetal death, neonatal death. Apgar score <7 at 5 minutes, birth weight <1500 g and <2500 g, use of mechanical ventilation, congenital anomaly.
Maternal Adverse events | up to 20 weeks from recruitment
  vaginal discharge, vaginal pruritus, discontinuation of treatment because of adverse events, threatened preterm labor.

REFERENCES:
- [Derived] Abdel-Aleem H, Shaaban OM, Abdel-Aleem MA, Aboelfadle Mohamed A. Cervical pessary for preventing preterm birth in singleton pregnancies. Cochrane Database Syst Rev. 2022 Dec 1;12(12):CD014508. doi: 10.1002/14651858.CD014508. PMID 36453699